CLINICAL TRIAL: NCT03449407
Title: Multi-dimensional Investigations of Negative Emotions and Drug-resistant Auditory Verbal Hallucinations in Psychosis
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Suzanne Ho-wai So, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: Mood&AVH
Record Dates: First submitted 2018-01-23; First posted 2018-02-28 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Schizophrenia Spectrum and Other Psychotic Disorders; Hallucinations, Auditory
Keywords: Auditory hallucinations; Psychosis; Mood; Brain imaging; Experience sampling method
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Hallucinations; Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Auditory verbal hallucinations (AVH) are commonly reported as source of distress, disability and mortality in schizophrenia. Despite proven efficacy of antipsychotics, many patients still experience drug-refractory AVH. It has been postulated that AVH is maintained by negative emotions. Yet, little is known about the temporal relationship and underlying mechanisms between negative affect and AVH. Utilizing both an ecologically-validated method and brain imaging technique, this study aims to uncover the role of emotions in the maintenance of psychotic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* Clinical diagnosis of schizophrenia spectrum disorder
* Present hallucinations

Exclusion Criteria:

* Left-handedness
* Intellectual disability
* Organic psychosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, including in-patients, out-patients and day hospital patients, will be recruited from psychiatric units of multiple hospital sites.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Psychotic symptomatology as measured by Positive and Negative Syndrome Scale (PANSS), Scale of Assessment for Positive Symptoms (SAPS), and the Psychotic Symptom Rating Scales (PSYRATS) | Baseline
  Positive and Negative Syndrome Scale (PANSS) is an interview-based assessment of the severity of symptoms associated with schizophrenia, including positive, negative, and general psychopathology. Scale of Assessment for Positive Symptoms (SAPS) is an interview-based scale of positive symptoms of schizophrenia. SAPS consists of four areas: hallucinations, delusions, bizarre behaviour and positive formal thought disorder. Each area includes ratings of specific symptoms and a global rating. The Psychotic Symptom Rating Scale (PSYRATS) is a 17-item semi-structured interview measuring the severity of multiple dimensions of auditory hallucinations and delusions, including conviction and duration.
Depressive symptomatology as measured by Calgary Depression Scale (CDS) | Baseline
  Calgary Depression Scale (CDS) is a nine-item structured interview scale that assesses depressive symptoms in patients with schizophrenia.
Beliefs about voices as measured by Beliefs about Voices Questionnaire - Revised (BAVQ-R) | Baseline
  BAVQ-R is a self-report questionnaire that consists of three subscales pertaining to beliefs about voices: malevolence (i.e. voices as evil and persecutory), benevolence (i.e. voices as helpful), and omnipotence (i.e. voices as controlling and powerful).
Anxiety severity as measured by Beck anxiety inventory (BAI) | 1 week
  BAI is a self-report questionnaire that measures anxiety severity and unique symptom features that are independent of that in depression, including somatic symptoms and subjective experience of panic and anxiety.
Mood states as measured by Visual analogue scale (VAS) | 1 week
  A simple visual analogue scale assessing state depression, state anxiety and state happiness will be conducted.

SECONDARY OUTCOMES:
Cognitive capacity as measured by the Wechsler Adult Intelligence Scale - IV (HK) short form (WAIS-IV) | Baseline
  An instrument developed to assess cognitive ability and the relationship between intellectual functioning and memory of adults. The WAIS-IV (HK) short form includes four subscales - arithmetic, visual puzzle, information, and coding.
Handedness as measured by Edinburgh Handedness Inventory (EHI) | Baseline
  A self report questionnaire assessing the dominance of one's right or left hand in everyday activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No